CLINICAL TRIAL: NCT00165958
Title: Comparison of Excision Versus Punch Incision in the Treatment of Epidermal Cysts
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Suephy Chen, MD, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1023-2004
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-07

CONDITIONS: Epidermal Cyst
Keywords: Epidermal cyst; Epidermoid cyst; Sebaceous cyst; Pilar cyst
MeSH Terms: conditions — Epidermal Cyst

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Punch excision (Experimental)
  Interventions: Procedure: Punch incision of epidermal cyst
- Traditional excision (Active Comparator)
  Interventions: Procedure: Excisional surgery of epidermal cyst

INTERVENTIONS:
Procedure: Excisional surgery of epidermal cyst — Traditional extirpation of cyst en toto
  Arms: Traditional excision
Procedure: Punch incision of epidermal cyst — removal of cyst first with incisional effort with a punch biopsy tool
  Arms: Punch excision

SUMMARY:
The purpose of this trial is to compare two standard of care treatments for removing epidermal cysts. Surgical excision removes the entire cyst but requires a larger hole in the skin. A punch incision makes a smaller hole through which the cyst can be removed. The trial's purpose is to determine if one method is better than another in terms of recurrence, infection, or other side effects.

DETAILED DESCRIPTION:
The purpose of this trial is to compare two standard of care treatments for removing epidermal cysts. Surgical excision removes the entire cyst but requires a larger hole in the skin. A punch incision makes a smaller hole through which the cyst can be removed. The trial's purpose is to determine if one method is better than another in terms of recurrence, infection, or other side effects.

Patients with epidermal cysts will be randomized to having the cyst removed by surgical excision or by a smaller punch incision followed by removal of the cyst through the smaller hole. The skin will be stitched shut in both cases. A short survey about how the cyst affects the patient will be given before the cyst is removed. When the stitches are removed 2 weeks later, photographs will be taken and a survey regarding satisfaction with the procedure will be given. Two additional phone surveys, given at 4 and 12 months after the procedure, wil be given to ask about recurrence, satisfaction with the procedure, side effects, and how the cyst affected the patient's life. The study doctor will be blinded as to which procedure each subject underwent. Forty subjects will be recruited at the Atlanta Veteran's Administration Medical Center

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years or older
* Epidermal cyst 1-3 cm in diameter on the trunk

Exclusion Criteria:

* Infected cyst requiring systemic antibiotics
* Pregnant females
* Unable to return to clinic for suture removal
* Previous excision of target cyst

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-01; Primary Completion 2008-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suephy C Chen, MD, Principal Investigator — Emory University Department of Dermatology
Locations (1):
- Atlanta VA Medical Center, Decatur, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: subjects older than 18 years of age with 1-3 cm truncal EICs were selected via serial recruitment from the Atlanta Veterans Affairs Medical Center Dermatology clinic
Pre-assignment Details: Patients were excluded if the cysts were inflamed, infected, or ruptured based on characteristic physical examination findings.
Groups:
- Punch Excision: Punch incision of epidermal cyst : removal of cyst first with incisional effort with a punch biopsy tool
- Traditional Excision: Excisional surgery of epidermal cyst : Traditional extirpation of cyst en toto
Period: Overall Study
Arm/Group | Punch Excision | Traditional Excision
Started | 19 | 21
Completed | 18 | 19
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Punch Excision | Traditional Excision | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 16 | 30
  >=65 years | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (11.8) | 59.0 (9.9) | 59.6 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 18 | 19 | 37
Region of Enrollment [Number; unit: participants]
  United States | 19 | 21 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Cyst Recurrence
Description: Recurrence of cyst after removal
Time Frame: 16 months
Measure: Number; unit: participants
Groups:
- Punch Incision: Punch incision of epidermal cyst : removal of cyst first with incisional effort with a punch biopsy tool
Arm/Group | Punch Incision | Traditional Excision
Number analyzed (Participants) | 19 | 17
participants | 3 | 2

ADVERSE EVENTS:
Arm/Group | Punch Incision | Traditional Excision
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 0/19 | 0/21

LIMITATIONS AND CAVEATS:
The limitations of this study include the small, predominately male patient population, lack of complete follow-up of secondary endpoint measurements at every time point.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No